CLINICAL TRIAL: NCT01330667
Title: Effect of Early Limited Formula on Total Serum Bilirubin Among Newborns With Hyperbilirubinemia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding not available
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ELF for Hyperbilirubinemia
Record Dates: First submitted 2011-02-23; First posted 2011-04-07 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Hyperbilirubinemia, Neonatal
Keywords: Hyperbilirubinemia; Breastfeeding; Limited Formula
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia; Breast Feeding | interventions — pregestimil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formula Supplementation (Experimental): Participants will supplement feedings with early limited formula following nursing.
  Interventions: Dietary Supplement: Nutramigen Infant Formula
- Control (No Intervention): Participants will be instructed to continue exclusively breastfeeding with no formula supplementation.

INTERVENTIONS:
Dietary Supplement: Nutramigen Infant Formula — Investigators will advise to supplement with 10cc's of extensively hydrolyzed formula immediately following each breastfeeding until TSB declines.
  Other Names: Nutramigen
  Arms: Formula Supplementation

SUMMARY:
The investigators propose to conduct an exploratory pilot study, enrolling 30 exclusively breastfeeding newborns 36-96 hours of age, whose Total Serum Bilirubin (TSB) is within 0.1-3 mg/dl of the American Academy of Pediatrics (AAP)-recommended treatment thresholds for Phototherapy (PT). These newborns will be randomly assigned to receive either 10 cc extensively hydrolyzed formula following each breastfeeding using cup, spoon or syringe, or to continue exclusive breastfeeding. Infants will be followed at 1, 2, 3 and 6 months to assess breastfeeding duration and use of formula and complementary foods. Our hypothesis is that limited, small amounts of formula administered without a bottle immediately following breastfeeding might reduce the incidence of severe hyperbilirubinemia among newborns at increased risk of TSB exceeding AAP-recommended thresholds for beginning phototherapy.

DETAILED DESCRIPTION:
Inclusion criteria

* Healthy infants ≥ 35 weeks
* Neonates 36-96 hours old
* Exclusively breastfeeding
* TSB 0.1-3 mg/dl below AAP-recommended PT threshold
* TSB < 6 hours ago
* Mothers English-speaking or Spanish-speaking

Outcome Measures

* Primary outcome: Total Serum Bilirubin
* Secondary clinical outcomes: Phototherapy, hospital readmission, exclusive and partial breastfeeding at 1 week, 1 month, 2 months, and 3 months; breastfeeding self-efficacy

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants ≥ 35 weeks
* Neonates 36-96 hours old
* Exclusively breastfeeding
* TSB 0.1-3 mg/dl below AAP-recommended PT threshold
* TSB < 6 hours ago
* Mothers English-speaking or Spanish-speaking

Exclusion Criteria:

* Infants who have already received formula
* Infants who have received or are receiving Level II or Level III
* Infants who have already lost ≥ 10% birth weight
* Infants with Glucose-6-phosphate dehydrogenase deficiency, positive direct antigen testing, cephalohematoma or other extensive bruising

Ages: 36 Hours to 96 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2015-07 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
TSB meeting or exceeding AAP-recommended phototherapy treatment threshold. | Up to two weeks after birth
  The investigators will compare measured TSB to AAP guideline recommendations for phototherapy treatment and confirming with Bili Tool, an automated program designed for this purpose.

SECONDARY OUTCOMES:
Receipt of phototherapy and hospital readmission, exclusive and partial breastfeeding at 1 week, 1 month, 2 months, and 3 months; breastfeeding self-efficacy | Up to three months after birth
  The investigators will ask mothers whether the infant received any breast milk in the last 24 hours. For infants whose mothers state they have received breast milk in the last 24 hours, the investigators will ask mothers whether the infant received anything other than breast milk in the last 24 hours. The investigators will ask mothers whether the infant received anything other than breast milk since the prior assessment. The investigators will query subjects using the Breastfeeding Self Efficacy Scale, short form, at enrollment, 1week and at 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Flaherman, MD,MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco Medical Center, San Francisco, California, United States